CLINICAL TRIAL: NCT06129630
Title: Effects of Nintendo Switch on Rehabilitation Programs for Elderly People With Cognitive Impairment: A Randomized Clinical Trial
Brief Title: Effects of Nintendo Switch on Rehabilitation Programs for Elderly People With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Cristina García-Bravo, PhD, Occupational Therapist, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2702202309423
Record Dates: First submitted 2023-10-30; First posted 2023-11-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Impairment; Elderly People; Healthy Aging; Occupational Therapy
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Control Group (CG), which received their usual sessions of conventional occupational therapy, and an Experimental Group (EG), which received therapy with Nintendo Switch, plus their conventional occupational therapy sessions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (Active Comparator): Control Group (CG), which received their usual sessions of conventional occupational therapy.
  Interventions: Procedure: Conventional occupational therapy sessions.
- Experimental Group (EG) (Experimental): Experimental Group (EG), which received therapy with Nintendo Switch, plus their conventional occupational therapy sessions.
  Interventions: Procedure: Conventional occupational therapy sessions + Nintendo Switch

INTERVENTIONS:
Procedure: Conventional occupational therapy sessions. — Occupational therapy sessions are based on cognitive stimulation, manipulative dexterity training and psychomotor skills.
  Arms: Control Group (CG)
Procedure: Conventional occupational therapy sessions + Nintendo Switch — Occupational therapy sessions are based on cognitive stimulation, manipulative skill training and psychomotor skills. In addition, 2 sessions per week are conducted with two Nintendo Switch games.
  Arms: Experimental Group (EG)

SUMMARY:
Purpose: Healthy aging is the process of optimizing opportunities for health, participation and safety in order to improve quality of life as people age. This study aimed to provide healthy aging for people with cognitive impairment through the use of the Nintendo Switch combined with Occupational Therapy sessions.

Material and methods: a randomized clinical trial was conducted. The sample was randomized using a software program, OxMar, which allowed the separation of the sample into a control group (CG), which received their usual sessions of conventional occupational therapy, and an experimental group (EG), which received therapy with Nintendo Switch, plus their conventional occupational therapy sessions. An 8-week intervention was conducted with Nintendo Switch.

Measures: Nine Hole Peg Test, Box and Block Test, Barthel Index, WHOQOL-BREF, CSQ-8.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women, aged 65 years or older, cohabitating in the nursing home.
* Not presenting moderate or severe cognitive impairment measured through the MEC- Lobo test (score ≥ 24-35) (20).
* Agree to participate voluntarily, having read the project information sheet and signed the informed consent.

Exclusion Criteria:

* Presence of neurodegenerative pathology.
* Presence of physical pathology that compromised the person's safety.
* Severe cognitive impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Nine Hole Peg Test | Pre-intervention and post-intervention (up to 1 week)
  This test measures fine manual dexterity. This is considered a "gold standard" to evaluate fine manual dexterity (21). It consists of placing a number of pins on a board with 9 holes and removing them as quickly as possible. This test records the time the person uses with each upper limb.
Box and Block Test | Pre-intervention and post-intervention (up to 1 week)
  Test that measures the gross motor skills of the upper limbs. It consists of a wooden box that is divided into two halves by an axis, and consists of passing from one half to the other as many wooden blocks as possible with each upper limb, for 1 minute. In this test, the number of blocks that the person is able to pass in one minute with each upper limb is recorded.
Barthel Index | Pre-intervention and post-intervention (up to 1 week)
  This scale is used to assess the level of functional independence in the basic activities of daily living that a person presents. In this test, the higher the score, the higher the level of functional independence of the person.
World Health Organization WHOQOL-BREF | Pre-intervention and post-intervention (up to 1 week)
  self-administered questionnaire, assesses the general perception of quality of life and general perception of health. It is composed of four domains: physical health, psychological health, social relationships and environment. A higher score on this scale indicates a higher quality of life. Potential scores for all domain scores, therefore, range from 4-20.

SECONDARY OUTCOMES:
The Client Satisfaction Questionnaire-8, CSQ-8 | Post-intervention (up to 1 week)
  Self-administered questionnaire used to evaluate satisfaction with the care services received, it consists of 8 questions. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction). Total scores range from 8 to 32, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Physiocare Madrid Clinic, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No